CLINICAL TRIAL: NCT06941350
Title: A Phase I/II Clinical Study Evaluating the Safety and Efficacy of NCR102 Injection in the Treatment of Acute Graft-versus-Host Disease (aGVHD)
Brief Title: A Trial to Evaluate the Safety and Efficacy of NCR102 in Subjects With aGVHD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nuwacell Biotechnologies Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCR102-1001
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Acute Graft-versus-Host Disease
Keywords: SR-aGVHD; NCR102; second-line treatment failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NCR102 injection (Experimental): Cohort1：Low dose NCR102 injection; Cohort2：High dose NCR102 injection
  Interventions: Biological: NCR102 injection

INTERVENTIONS:
Biological: NCR102 injection — Twice a week for 4 weeks, and the treatment continues for another 4 weeks in subjects with partial remission by day 28.

SUMMARY:
Evaluate the safety and efficacy of NCR102 injection in the treatment of SR-aGVHD patients who have failed second-line therapy.

DETAILED DESCRIPTION:
An open-label, dose-escalation and dose-expansion study to evaluate the safety, tolerability and preliminary efficacy of NCR102 injection in the treatment of SR-aGVHD patients who have failed second-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years and <70 years old (including threshold), gender not limited；
* Grade II to IV gastrointestinal involvement acute graft-versus-host disease(aGVHD)；
* Subjects with Steroid-refractory Acute Graft-versus-host Disease(SR-aGVHD)；
* Failed to second-line aGVHD treatment;
* Subjects will receive NCR102 injection treatment within 3 days after enrollment;
* Voluntarily sign an informed consent form.

Exclusion Criteria:

* Subjects have lung disease, and investigators have determined that they are not suitable for the study;
* Subjects with severe hepatic vein occlusion disease or sinus vein occlusion syndrome;
* Subjects with signs/symptoms of chronic GVHD;
* Subjects who are clinically assessed by the investigator could not be ruled out as having diarrhea caused by cytomegalovirus (CMV) enteritis, transplant related thrombotic microvascular disease (TA-TMA), or digestive tract infection;
* Eastern Cooperative Oncology Group(ECOG)>3；
* Subjects have other diseases or physiological conditions that may interfere with the evaluation results of this trial, or life-threatening complications；
* Subjects had active malignant solid tumors within the past 5 years；
* Subjects had a known history of severe allergies to blood products, or heterologous proteins.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Event(AE) or Serious Adverse Event(SAE) | 100 days after first administration of NCR102 injection
  Number of participants with treatment-related adverse events or serious adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
ORR at Day 28 | 28 days after first dose administration
  Overall Response Rate(ORR) at Day 28
CRR at Day 28 | 28 days after first dose administration
  Complete Response Rate(CRR) at Day 28
ORR at Day 56 | 56 days after first dose administration
  Overall Response Rate(ORR) at Day 56